CLINICAL TRIAL: NCT06249126
Title: Primary Subtalar Arthrodesis for Calcaneal Fractures to Optimize Performance: A Randomized Clinical Trial
Brief Title: Primary Subtalar Arthrodesis for Calcaneal Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00107954; HT94252310505 (Other: Department of Defense)
Record Dates: First submitted 2024-01-30; First posted 2024-02-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-06

CONDITIONS: Calcaneus Fracture
Keywords: heel injuries; post-traumatic subtalar arthritis; orthopaedic injury
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Fusion (Open Reduction Internal Fixation (ORIF) + Primary Subtalar Arthrodesis (PSTA) (Other): Surgical fixation by joint fusion + Surgical fixation with plates and screws, plates, sutures, or rods are used to hold the broken bone together
  Interventions: Procedure: Primary Fusion (Open Reduction Internal Fixation (ORIF) + Primary Subtalar Arthrodesis (PSTA)
- Open Reduction Internal Fixation (ORIF) only (Other): Surgical fixation with plates and screws, plates, sutures, or rods are used to hold the broken bone together
  Interventions: Procedure: Open Reduction Internal Fixation (ORIF) only

INTERVENTIONS:
Procedure: Primary Fusion (Open Reduction Internal Fixation (ORIF) + Primary Subtalar Arthrodesis (PSTA) — Definitive fixation by joint fusion
  Arms: Primary Fusion (Open Reduction Internal Fixation (ORIF) + Primary Subtalar Arthrodesis (PSTA)
Procedure: Open Reduction Internal Fixation (ORIF) only — Definitive fixation with plates and screws
  Arms: Open Reduction Internal Fixation (ORIF) only

SUMMARY:
Management of severe injuries to the heel (displaced intra-articular calcaneus fractures) continues to be a major challenge for orthopedic surgeons. Previous studies have demonstrated poor outcomes, and results show that patients experience long-term pain and decreased quality of life postoperatively. Poor outcomes are driven by pain, in particular, which is linked to post-traumatic subtalar arthritis.

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare two surgical options for calcaneus fractures to determine best treatment for returning to work sooner in adults.

Participants will be randomized to one of two treatment options and will be asked to complete patient reported outcome measure surveys.

Researchers will compare Open Reduction and Internal Fixation (ORIF) + Primary Subtalar Arthrodesis (PSTA) to ORIF alone to see which group returns to work at an earlier timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing operative treatment for displaced intra-articular calcaneus fracture
* Sanders III and IV displaced intra-articular calcaneus fracture OR Sanders II with any of the following criteria: Bohler angle < 0 degrees, open fracture, pain syndrome, substance use disorder
* Age 18 or older
* Able to follow up at site for 1 year

Exclusion Criteria:

* Planned surgery using extensile lateral approach
* Sanders II displaced intra-articular calcaneus fracture without: Bohler angle < 0 degrees, open fracture, pain syndrome, or substance
* <18 years of age
* Body Mass Index (BMI) >40
* Unable to follow up at site for 1 year
* Patients that speak neither English or Spanish
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Return to Work/Duty - Metabolic Equivalent for Tasks (METs) Score | Week 6
  The primary outcome is return to work/duty as measured by the International Physical Activity Questionnaire (IPAQ). The IPAQ is a validated, self-report measure that captures detailed information about participation in a wide range of physical activities, including the number of days and amount of time spent in the previous 7 days. Responses for each type of physical activity are then transformed into the number of Metabolic Equivalent for Tasks (METs), and a METs/week is calculated for each patient. The IPAQ has moderate concordance with accelerometry-measured METs in an orthopaedic injury patient population.
  (one MET is defined as 3.5 mL O2 uptake/kg per min, which is the resting oxygen uptake in a sitting position). Less than 5 METS is poor, 5-8 METS is fair, 9-11 METS is good, and 12 METS or more is excellent.
Return to Work/Duty - Metabolic Equivalent for Tasks (METs) Score | Week 12
  The primary outcome is return to work/duty as measured by the International Physical Activity Questionnaire (IPAQ). The IPAQ is a validated, self-report measure that captures detailed information about participation in a wide range of physical activities, including the number of days and amount of time spent in the previous 7 days. Responses for each type of physical activity are then transformed into the number of Metabolic Equivalent for Tasks (METs), and a METs/week is calculated for each patient. The IPAQ has moderate concordance with accelerometry-measured METs in an orthopaedic injury patient population.
  (one MET is defined as 3.5 mL O2 uptake/kg per min, which is the resting oxygen uptake in a sitting position). Less than 5 METS is poor, 5-8 METS is fair, 9-11 METS is good, and 12 METS or more is excellent.
Return to Work/Duty - Metabolic Equivalent for Tasks (METs) Score | Month 6
  The primary outcome is return to work/duty as measured by the International Physical Activity Questionnaire (IPAQ). The IPAQ is a validated, self-report measure that captures detailed information about participation in a wide range of physical activities, including the number of days and amount of time spent in the previous 7 days. Responses for each type of physical activity are then transformed into the number of Metabolic Equivalent for Tasks (METs), and a METs/week is calculated for each patient. The IPAQ has moderate concordance with accelerometry-measured METs in an orthopaedic injury patient population.
  (one MET is defined as 3.5 mL O2 uptake/kg per min, which is the resting oxygen uptake in a sitting position). Less than 5 METS is poor, 5-8 METS is fair, 9-11 METS is good, and 12 METS or more is excellent.
Return to Work/Duty - Metabolic Equivalent for Tasks (METs) Score | Month 12
  The primary outcome is return to work/duty as measured by the International Physical Activity Questionnaire (IPAQ). The IPAQ is a validated, self-report measure that captures detailed information about participation in a wide range of physical activities, including the number of days and amount of time spent in the previous 7 days. Responses for each type of physical activity are then transformed into the number of Metabolic Equivalent for Tasks (METs), and a METs/week is calculated for each patient. The IPAQ has moderate concordance with accelerometry-measured METs in an orthopaedic injury patient population.
  (one MET is defined as 3.5 mL O2 uptake/kg per min, which is the resting oxygen uptake in a sitting position). Less than 5 METS is poor, 5-8 METS is fair, 9-11 METS is good, and 12 METS or more is excellent.

SECONDARY OUTCOMES:
Number of Complications | Week 6, Months 3 and 6
  Major complications, including infection, nonunion, malunion, and hardware failure will be captured from the medical record.
Number of Return to Operating Room Visits | Week 6, Months 3 and 6
  Details regarding reoperations will be collected, especially in cases of hardware removal and those randomized to Open Reduction Internal Fixation (ORIF) who receive secondary subtalar fusion.
Number of Resource Utilizations | Week 6, Months 3 and 6
  Healthcare utilization, including new hospitalizations, emergency department visits, clinic visits, imaging, and physical therapy sessions will be documented at all follow-up visits
Rates of Symptomatic Arthritis - Kellgren Lawrence (KL) classification | 1 year
  If post-traumatic osteoarthritis (PTOA) is present, Kellgren Lawrence (KL) classification (This semiquantitative approach primarily evaluates osteophytes and joint space narrowing to assign a score between 0 (no ROA) to 4 (severe ROA) will be assessed by the panel of reviewers and documented.
Rates of Symptomatic Arthritis - Paley Grading System (PGS) | 1 year
  If post-traumatic osteoarthritis (PTOA) is present, the Paley Grading System (PGS) will be assessed by the panel of reviewers and documented - type 1: tibial shortening alone with a normal ankle (A); type 2: tibial shortening with dynamic valgus at the ankle (B)
Current Pain Level Ratings | Week 6, Months 3 and 6 and 12
  Pain will be assessed using the Numeric Rating Scale. Patients will be asked to rate their current pain at each visit. Patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Union | 1 year
  Union, as determined by the treating surgeon, will be assessed via radiographs and documented as a dichotomous outcome (yes/no), and time to union will also be captured. Nonunion will be captured via surgeon diagnosis or return to the operating room for nonunion treatment.
Patient-Reported Outcomes Measurement Information System (PROMIS) 29 Scores | Week 6, Months 3 and 6 and 12
  The PROMIS-29 is a free to use, publicly available generic health related quality of life measure that includes seven domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities. A 5-point Likert scale is used for each question and norm-based total scores (range 0-100) have been calculated so that 50 represents the mean and one standard deviation is 10 points. Additionally, higher scores represent better function.
Veterans RAND 12 Item Health Survey (VR-12) Scores | Week 6, Months 3 and 6 and 12
  The VR-12 is a measure of global health that correspond to seven domains: general health, physical functioning, role limitations, pain, fatigue, social functioning, and mental health. Together, these items are summarized into a Physical Component Score and a Mental Component Score. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Work Productivity and Activity Impairment Questionnaire Scores | Week 6, Months 3 and 6 and 12
  If return to duty/work is reported, patients will complete the Work Productivity and Activity Impairment Questionnaire, a validated instrument that measures work time missed and work and activity impairment due to health problems. Measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. The higher number of day equates to more health problems
Tampa Scale for Kinesiophobia (TSK) Scores | Week 6, Months 3 and 6 and 12
  This scale is 17 items and uses a 4-point Likert scale ranging from 'strongly disagree' to 'strongly agree'. The TSK is a validated measure for surgical and musculoskeletal patients. The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia
Counter-Movement Jump - Height | Upon being cleared for high level activity, Week 6, Months 3 and 6 and 12
  Patients will be asked to perform a double-leg and single-leg countermovement jump to assess jump height. Patients will be asked to perform three repetitions of countermovement jump for maximal height off of a force plate followed by landing on the same force plate. The average jump height (centimeters),will be calculated across the three trials.
Counter-Movement Jump - force development (percent body weight/milliseconds) | Upon being cleared for high level activity, Week 6, Months 3 and 6 and 12
  Patients will be asked to perform a double-leg and single-leg countermovement jump to assess concentric force development (take-off) (VALD Force Deck System). Patients will be asked to perform three repetitions of countermovement jump for force development (percent body weight/milliseconds) and will be calculated across the three trials.
Counter-Movement Jump - force dissipation (percent body weight/milliseconds) | Upon being cleared for high level activity, Week 6, Months 3 and 6 and 12
  Patients will be asked to perform a double-leg and single-leg countermovement jump to assess force dissipation (landing) (VALD Force Deck System). Patients will be asked to perform three repetitions of countermovement jump for maximal height off of a force plate followed by landing on the same force plate. The average jump force dissipation (percent body weight/milliseconds) will be calculated across the three trials.
Single Leg Static Percentage | Upon being cleared for high level activity, Week 6, Months 3 and 6 and 12
  Static postural stability will be assessed under eyes open and eyes closed conditions. The average of three 10-second trials will be collected for data analysis for each condition. The variable to be analyzed will the standard deviation of resultant ground reaction force across the 10-second trial. It will be a percentage.
Dynamic Postural Stability Percentage | Upon being cleared for high level activity, Week 6, Months 3 and 6 and 12
  Dynamic postural stability will be assessed during a single-leg landing. Patients will be asked to jump forward to the force plate, clear a 30.5 cm hurdle, land on the force plate with their test leg only, stabilize as quickly as possible, and maintain balance with their hands on their hips for ten seconds. A total of three trials will be collected and averaged together for analysis. A stability index based on the three ground reaction force components will be calculated. The unit of Force will be in percent body weight. It will be a percentage. The higher the percentage, indicating better stability.
Triple Hop Performance Assessment Length | Upon being cleared for high level activity, Week 6, Months 3 and 6 and 12
  Bilateral assessment of jump performance will be performed during a triple hop (cross-over) for maximum distance. Participants will be provided a practice trial at 50 percent maximum effort prior to the test trials and testing will begin with non-surgical left first. Participants will begin the jump behind zero-inch line, which marks the starting point. Participants will perform three consecutive jumps off one leg while crossing over the tape with each jump so that the first jump is lateral, the second jump is medial, and the final jump is lateral. Participants will be asked to hold their place at the end of the third jump until their distance is recorded. Three test trials will be assessed for each leg and averaged together for analysis.
Pain Intensity Scores | Week 6, Months 3 and 6 and 12
  Pain will be assessed using the Brief Pain Inventory (BPI). The BPI is a commonly used and validated 15-item measure of pain intensity and interference with daily life. Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Pain Interference Scores | Week 6, Months 3 and 6 and 12
  Pain will be measured with the pain intensity and pain interference Patient-Reported Outcomes Measurement Information System (PROMIS) domains. Score on a scale from 0 to 100, where higher Pain Intensity and Pain Interference scores indicate inferior outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Hsu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (14):
- United States (14):
  - Emory University, Grady Memorial Research Hospital, Atlanta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University - University Medical Center New Orleans, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - NYC Health and Hospital/Bellevue, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - OrthoCarolina Foot and Ankle Institute, Charlotte, North Carolina
  - Atrium Health Cabarrus, Concord, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Prisma Health, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No